CLINICAL TRIAL: NCT04055103
Title: Improving Quality Based on the Joint Registry
Acronym: IQ Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, PerlaJMarang, Associate Professor, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: G18.140; VRF2018-001 (Other Grant/Funding Number: Van Rens Foundation)
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Registries; Quality Improvement; Hip Arthropathy; Knee Arthropathy; Hospital Performance
Keywords: Total Hip/Knee Arthroplasty;Dutch Arthroplasty Register; Quality Improvement.
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Each arm will receive the intervention for 6 months.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Half of the participating hospitals will be in the intervention group for the first 6 months. The intervention will switch to the control group after the 6 months.
  Interventions: Other: Monthly feedback, education and linking hospitals
- Control Group (No Intervention): Half of the participating hospitals will be in the control group for the first 6 months. The control group will undergo the intervention in the second 6 months.

INTERVENTIONS:
Other: Monthly feedback, education and linking hospitals — - Give monthly feedback from LROI-data (revision rate & patient reported outcome measures) as well as other outcomes from the participating hospital (length-of-stay, readmission and complications), combined with education on how to use this information for improvement. This will be send monthly by email to the intervention group. Further, hospitals with worse performance for a certain outcome will be linked to hospitals with good performance for this outcome.
  Arms: Intervention Group

SUMMARY:
Test whether an intervention, consisting of frequently feedback of performance outcomes and education will improve patient care, expressed in better functional outcomes, fewer complications and more quality improving interventions.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted where hospitals will be randomized to an early versus late group, stratified by teaching status as this might influence the time available for quality improvement. Randomization will be done using a computer generated randomization table in a 1:1 ratio. During the study only orthopedic surgeons performing THA and TKA will receive monthly feedback by email.

The intervention will consist of the following components:

* Monthly feedback of performance outcomes;
* Education on how to use joint registry data for quality improvement;
* Create awareness by sending monthly feedback about performance; education and by asking what improvement activities have been introduced;
* Hospitals will be linked to hospital with opposite performance outcomes to exchange information and find areas for improvement.

During the trial, the investigators will conduct monthly measurement on intermediate outcomes showing whether the intervention reaches the target group (process evaluation). The following measurements will take place:

* Knowledge among orthopaedic surgeons on their recent performance and how that relates to others;
* Number of quality improvement activities undertaken with the aim to improve the quality of care;
* Planned improvement activities (e.g. record review to figure out why performance is not as good as in other centers) together with who is responsible and by which time;
* Number of people attending the meetings, number of times a specific account has accessed the LROI site to ensure that information has reached the target group;
* Survey among orthopaedic surgeons at the end of the intervention period on knowledge learned and the extent to which they think this is sustainable in daily practice.

In addition, the investigators will compare the outcomes between the early and the late group to test the effectiveness of the intervention, using the appropriate regression techniques. In the second period the investigators will test the sustainability of this approach in daily practice by comparing the outcomes within the early group with the first period, and compare with the late group to test whether outcomes in the sustainability phase are similar as when actively supported.

ELIGIBILITY:
Inclusion Criteria:

* All Dutch orthopedic clinics where hip- and knee replacement surgery is performed who agree to participate will be randomized.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Survival (yes/no) | 1 year follow-up during trial
  Patient survival after HA/TKA surgery
1-year revision rate (%) | 1 year follow-up during trial
  Number of revisions performed within one year adjusted for patient characteristics
Prolonged length-of stay (yes/no) | 1 year follow-up during trial
  Prolonged length-of-stay in the overall upper quartile
Readmission (yes/no) | 1 year follow-up during trial
  Readmission within 30 days after discharge
Number of Complications | 1 year follow-up during trial
  Number of complications
Composite outcome measure (Textbook Outcome) | 1 year follow-up during trial
  Including: Survival; 1-year revision rate; Length-of-Stay and Readmission.

SECONDARY OUTCOMES:
Number of Quality Improvement Initiatives | 1 year follow-up during trial
  Number of quality improvement Initiatives with the aim to improve the quality of care

CONTACTS AND LOCATIONS:
Overall Officials: Perla Marang-van de Mheen, Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
This is about the performance of hospitals. The individual performance of a hospital will not be announced.

REFERENCES:
- [Derived] van Schie P, van Bodegom-Vos L, Zijdeman TM, Nelissen RGHH, Marang-van de Mheen PJ; IQ Joint study group. Effectiveness of a multifaceted quality improvement intervention to improve patient outcomes after total hip and knee arthroplasty: a registry nested cluster randomised controlled trial. BMJ Qual Saf. 2023 Jan;32(1):34-46. doi: 10.1136/bmjqs-2021-014472. Epub 2022 Jun 22. PMID 35732486

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Main protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04055103/Prot_SAP_000.pdf
  • Study Protocol: Annex 1: Grant Application Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04055103/Prot_001.pdf
  • Study Protocol: Annex 2: Data Delivery Agreement (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04055103/Prot_002.pdf